CLINICAL TRIAL: NCT01177475
Title: Effect of Intake in Bioactive Molecules From Natural or Pasteurised Milk on Gut Maturation in Very Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-A00666-51; 2009 09 (Other: AP HM)
Record Dates: First submitted 2010-03-18; First posted 2010-08-09 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Premature Birth
Keywords: kidney-transplant recipients
MeSH Terms: conditions — Premature Birth | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- natural milk (Active Comparator)
  Interventions: Other: blood samples, feces samples
- pasteurized milk (Experimental)
  Interventions: Other: blood samples , feces samples

INTERVENTIONS:
Other: blood samples , feces samples — After the 32nd week until the 36th week or the end of hospitalization,infants received mother's native milk or substitute.
  Arms: pasteurized milk
Other: blood samples, feces samples — After the 32nd week until the 36th week or the end of hospitalization,infants continued mother's native milk or received substitute.
  Arms: natural milk

SUMMARY:
It seems important to correlate real consumption in bioactives molecules of natural milk versus pasteurized with gut maturation in very preterm infants during small enteral feeding protocol. This objective will be reached through a clinical trial.

DETAILED DESCRIPTION:
One hundred infants born between 28 and 30 weeks of gestational age will be enrolled in our clinical trial in two neonatal units of Marseille; they will receive small enteral feeding protocol with natural or pasteurized milk (according to the Neonatology Department). Infants monitoring will be conducted from birth until 32 weeks of gestational age through extra-uterine growth, dietary type evolution and determination of gut maturation markers levels in blood (Triglycerides and Cholesterol, PUFA, GLP-2, I and L-FABP, Gastrin, Citrullin) and faeces (Calprotectine). We will also look for new biological markers of intestinal growth, via metabolomic approach. Consumption of bioactives molecules (PUFA, sphingomyelin, sCD14, insulin, leptin, lactoferrin, sphingomyelinase acid and BSSL activity) will be quantified in milk 24h-representative samples received by each newborn. The benefits on digestive tract physiology evolution due to the molecules consumption will be observed from the 32nd week until the 36th week or the end of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Children whose term is understood(included) between 28 (27SA+6j past(over)) and 30 LIMITED COMPANIES (30 SA+6j).
* Children fed by digestive stimulation.
* Children in 1st day of food(supply)
* Term of certain child.
* Children not presenting a genic syndrome, an evolutionary neurological disease, a pathology malformative.
* Children among whom both holders of the parental authority are of more than 18 years old and are not major protected by the law or deprived of freedom.
* Children among whom the relatives(parents) or the legal representatives accepted the participation of their child in this study, and having signed a lit(enlightened) consent.

Exclusion Criteria:

* Children been born > 30 LIMITED COMPANIES and < 28 limited companies.
* Children presenting a genic syndrome, an evolutionary neurological disease, a pathology malformative.
* Children among whom the relatives(parents) or the legal representatives refused that their child participates in the study.

Ages: 1 Day to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pasteurized milk | 2 years
  infants born between 28 and 30 weeks of gestational age will receive small enteral feeding protocol with pasteurized milk

SECONDARY OUTCOMES:
natural milk | 2 years
  infants born between 28 and 30 weeks of gestational age will receive small enteral feeding protocol with natural milk

CONTACTS AND LOCATIONS:
Overall Officials: CATHERINE GIRE, Principal Investigator — ASSITANCE PUBLIQUE HOPITAUX DE MARSEILLE; CATHERINE GIRE, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France